CLINICAL TRIAL: NCT06578390
Title: Efficacy Investigation of the Medical Device Apneal® on Smartphone for Sleep Apnea-Hypopnea Syndrome Diagnosis
Acronym: SESAME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mitral (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-A00042-45
Record Dates: First submitted 2024-08-21; First posted 2024-08-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Sleep Apnea Syndromes
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Each patient will wear the device and polysomnograph at the same time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Patients will wear the device during their polysomnographic recording
  Interventions: Device: Apneal device

INTERVENTIONS:
Device: Apneal device — Patients will wear a smartphone with the Apneal Application on their chest, while they perform polysomnography

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the Apneal® app in diagnosing sleep apnea syndrome (SAS) in adults who require polysomnography (PSG) as part of routine care. The main questions it aims to answer are:

* Can Apneal® accurately classify the SAS severity into four categories (normal: AHI < 5, mild: 5 ≤ AHI < 15, moderate: 15 ≤ AHI < 30, and severe: AHI ≥ 30) compared to PSG ?
* How does Apneal® perform in estimating the Apnea-Hypopnea Index (AHI), detecting sleep stages, differentiating between central and obstructive apneas, and identifying patient movements?

Participants will:

* Wear the Apneal® app-equipped smartphone and undergo PSG during a full night of sleep at home.
* Complete several questionnaires assessing sleep symptoms and experience with the Apneal® app.

ELIGIBILITY:
Inclusion Criteria:

* Individuals, male or female, aged 18 years or older (no upper age limit).
* Individuals for whom polysomnography (PSG) is indicated as part of routine care, regardless of the specific indication.
* Individuals with a reported total sleep time of at least 6 hours, in accordance with AASM recommendations for PSG analysis.
* Individuals affiliated with social security or benefiting from a similar system, if applicable, in accordance with local regulations.
* Voluntary individuals who have provided oral and written consent after being informed by the research investigator.

Exclusion Criteria:

* Individuals with an active implantable medical device (e.g., electronic cardiac implant, neurophysiological electrical stimulator).
* Individuals with a chest deformity that prevents proper placement of the smartphone on the chest.
* Individuals with uncontrolled psychiatric disorders that prevent them from giving full consent to the study.
* Individuals unable to understand or speak the official language of the research center.
* Individuals currently excluded from another protocol or participating in another interventional research study.
* Vulnerable persons or adults under legal protection, including pregnant or breastfeeding women, persons deprived of liberty by judicial or administrative decision, individuals hospitalized without consent, or admitted for purposes other than research (Articles L1121-5 to L1121-8 of the French Public Health Code).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate the performance of Apneal® in diagnosing sleep apnea-hypopnea syndrome (SAHS) | through study completion, an average of 1 year
  Performance of Apneal® in classifying the severity of SAHS into four categories (normal: AHI < 5, mild: 5 ≤ AHI < 15, moderate: 15 ≤ AHI < 30, severe: AHI ≥ 30) compared to polysomnography (PSG).

SECONDARY OUTCOMES:
Estimate the Apnea-Hypopnea Index (AHI) using Apneal® | through study completion, an average of 1 year
  Concordance of AHI measured by Apneal® with AHI measured by PSG, and the mean absolute error between the two measurements.
Compare Apneal® with screening questionnaires (NoSAS, Berlin, Epworth) | through study completion, an average of 1 year
  Comparison of Apneal®'s performance with the NoSAS, Berlin, and Epworth questionnaires in classifying the severity of SAHS into the four categories (normal, mild, moderate, severe) relative to PSG.
Detect sleep stages using Apneal® | through study completion, an average of 1 year
  The minimum concordance between Apneal® and PSG for both sleep stage durations (wake, REM, NREM: N1, N2, N3) and sleep stage latencies.
Differentiate central and obstructive apneas using Apneal® | through study completion, an average of 1 year
  Estimation of the Central Apnea Index (CAI) by Apneal® compared to PSG, indicating the number of central apneas per hour of sleep.
Detect patient movements with Apneal® | through study completion, an average of 1 year
  Comparison of night segmentation by movements (presence/absence) between Apneal® and PSG, and evaluation of the number of movements detected by both.
Evaluate patient acceptability of Apneal® | through study completion, an average of 1 year
  Percentage of patients who agree to participate vs. those who refuse, including reasons for refusal (e.g., equipment-related issues, cognitive impairment).
Assess the feasibility of SAHS screening using Apneal® | through study completion, an average of 1 year
  Percentage of patients with usable data provided by Apneal® out of the total number of patients included; data considered unusable if Apneal® is lost during the night.

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Wanono, MD, Principal Investigator — CHU de Reims
Locations (11):
- France (11):
  - Centre de pneumologie et sommeil, Aix-en-Provence
  - Centre du sommeil d'Antony, Antony
  - Pôle d'Exploration des Apnées du Sommeil de la Nouvelle Clinique Bel-Air, Bordeaux
  - SomnoLab - Millénaire, Montpellier
  - Cabinet de médecine du sommeil - Cabsom, Mulhouse
  - Somnology, Paris
  - Institut médical du sommeil, Paris
  - Cabinet privé du Dr. Wanono, Reims
  - Clinique du Renaison, Roanne
  - Somnidoc, Roanne
  - Centre Clinical, Soyaux

IPD SHARING:
Plan to Share IPD: No